CLINICAL TRIAL: NCT03954119
Title: Prognostic Relevance of Elevated Blood Pressure in the Emergency Department
Brief Title: Blood Pressure in the Emergency Department
Acronym: PREBPED
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Svensson, Associate professor, Karolinska Institutet
Other Study IDs: BPED1605
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Blood Pressure; Hypertension; Emergencies
Keywords: blood pressure; emergency department; atherosclerotic cardiovascular disease; myocardial infarction; stroke; long-term prognosis
MeSH Terms: conditions — Hypertension; Emergencies; Atherosclerosis; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cohort study based on a large sample (> 600 000) of emergency department (ED) visits from two university hospital EDs. Information on incident disease after discharge from the ED will be collected through linkage to Swedish national in-patient register and cause of death register. The importance of blood pressure measured at the ED for incident atherosclerotic cardiovascular disease during long term follow up will be studied by Cox-regression analysis

ELIGIBILITY:
Inclusion Criteria:

* Attending the Emergency departments (ED) at Karolinska University hospital in Solna or Huddinge during the specified time period
* Record of blood pressure measurement from the ED-visit

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected adult patients attending the ED irrespective of chief complaint
Sampling Method: Non-Probability Sample
Enrollment: 300272 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Incident Atherosclerotic Cardiovascular Disease (ASCVD) | 20161231
  ASCVD was defined as a combination of fatal coronary heart disease (CHD ), (I210-I214, I219, I220, I221, I228, I229, I461 or I469), non-fatal MI (I210-I214, I219, I220, I221, I228 or I229), fatal and non-fatal ischemic stroke (I630-I635, I638 or I639). According to the International Classification of Diseases 10th edition (ICD-10).

SECONDARY OUTCOMES:
Incident Myocardial infarction (MI) | 2016-12-31
  Fatal and non-fatal Myocardial infarction (MI) I210-I214, I219, I220, I221, I228 or I229. I200 were included if combined with intervention procedure codes FNA-FNG, FNW) , according to the International Classification of Diseases 10th edition (ICD-10).
Incident All-cause stroke | 2016-12-31
  Fatal and non-fatal all-cause stroke. I61, I630-I635, I638, I639, I64, according to the International Classification of Diseases 10th edition (ICD-10).
Incident Heart failure | 2016-12-31
  I50 according to the International Classification of Diseases 10th edition (ICD-10).
Incident chronic kidney disease (CKD) | 2016-12-31
  I120, I131 E10.2-E10.5,E10.7,E11.2-E11.5, E11.7,E12.2-E12.5,E12.7, E13.2- E13.5,E13.7,E14.2-E14.5, E14.7 N032-037, N052-057, N18, N19, N250, Z49,Z49.0,Z49.1, Z49.2,Z49.01, Z49.02,Z49.3,Z49.31,Z49.32, Z99.2, I77.0 Z94.0 according to the International Classification of Diseases 10th edition (ICD-10).

CONTACTS AND LOCATIONS:
Overall Officials: Per O Svensson, MD PhD, Principal Investigator — Department of Clinical Science and Education, Södersjukhuset |

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oras P, Habel H, Skoglund PH, Svensson P. Elevated Blood Pressure in the Emergency Department: A Risk Factor for Incident Cardiovascular Disease. Hypertension. 2020 Jan;75(1):229-236. doi: 10.1161/HYPERTENSIONAHA.119.14002. Epub 2019 Dec 2. PMID 31786971